CLINICAL TRIAL: NCT01796691
Title: Optimized Antiplatelet Therapy With Aspirin and Clopidogrel Improves Mortality Compared to Standard Treatment.
Brief Title: The Bochum Optimizing Clopidogrel-Aspirin Therapy and MORTality Study (BOCLA-Mort)
Acronym: BOCLA-Mort
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Horst Neubauer, PHD, MD, Ruhr University of Bochum
Other Study IDs: BOCLAplan02; [Ruhr-University Bochum] (Registry Identifier: F654R)
Record Dates: First submitted 2013-02-17; First posted 2013-02-22 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Artery Disease
Keywords: Clopidogrel; aspirin; low response; platelet aggregation; Acute Coronary Syndrome; Coronary Stent Implantation
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard therapy: Antiplatelet therapy following coronary stenting without platelet function testing
- Optimized antiplatelet therapy: Platelet function testing and according to a test and treat strategy improve the antiplatelet therapy in low-responder.
  Treatment adjustments were done as published before - see BOCLA-Plan manuscript. (Reference: Tailored antiplatelet therapy can overcome clopidogrel and aspirin resistance--the BOchum CLopidogrel and Aspirin Plan (BOCLA-Plan) to improve antiplatelet therapy. BMC Med. 2011 Jan 12;9:3.)

SUMMARY:
Comparing standard treatment versus optimized antiplatelet therapy and outcomes measures.

DETAILED DESCRIPTION:
The study is aimed to evaluate if optimized antiplatelet treatment using a test and treat algorithm (with whole blood aggregometry) is able to improve clinical outcome of patients compared to standard treatment without platelet function testing.

ELIGIBILITY:
Inclusion Criteria:

* coronary stent implantation

Exclusion Criteria:

* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients following coronary stenting if informed consent was obtained
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2009-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Adverse cardiac events (MACE: mortality,rehospitalisation,myocardial infarction) | Follow up for up to 12 months (retrospective analysis)
  MACE-rate

CONTACTS AND LOCATIONS:
Overall Officials: Horst Neubauer, MD, Principal Investigator — Ruhr-University Bochum, Cardiovascular Center
Locations (1):
- Cardiovascular Center, Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Neubauer H, Kaiser AF, Endres HG, Kruger JC, Engelhardt A, Lask S, Pepinghege F, Kusber A, Mugge A. Tailored antiplatelet therapy can overcome clopidogrel and aspirin resistance--the BOchum CLopidogrel and Aspirin Plan (BOCLA-Plan) to improve antiplatelet therapy. BMC Med. 2011 Jan 12;9:3. doi: 10.1186/1741-7015-9-3. PMID 21226927
- [Background] Neubauer H, Lask S, Engelhardt A, Mugge A. How to optimise clopidogrel therapy? Reducing the low-response incidence by aggregometry-guided therapy modification. Thromb Haemost. 2008 Feb;99(2):357-62. doi: 10.1160/TH07-10-0624. PMID 18278186
- [Background] Siller-Matula JM, Francesconi M, Dechant C, Jilma B, Maurer G, Delle-Karth G, Gouya G, Ruzicka K, Podczeck-Schweighofer A, Christ G. Personalized antiplatelet treatment after percutaneous coronary intervention: the MADONNA study. Int J Cardiol. 2013 Sep 1;167(5):2018-23. doi: 10.1016/j.ijcard.2012.05.040. Epub 2012 May 30. PMID 22656044